CLINICAL TRIAL: NCT01110200
Title: A Randomized, Double-Blind, Parallel Group, Multicenter Study of the Effects of Fluticasone Propionate/Salmeterol Combination Product 250/50mcg BID (ADVAIR DISKUS™) in Comparison to Salmeterol 50mcg BID (SEREVENT DISKUS™) on the Rate of Exacerbations of COPD Following Hospitalization
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) Post-hospitalization Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113874
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Hospitalization; Exacerbations of COPD; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination; BID protein, human; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADVAIR DISKUS 250/50 mcg BID (Active Comparator): Fluticasone propionate/salmeterol 250/50 mcg BID in the DISKUS formulation (ADVAIR DISKUS) is a combination product containing a corticosteroid and a long-acting beta2-adrenergic agonist, indicated in the US for the maintenance treatment of airflow obstruction and reducing exacerbations in patients with COPD.
  Interventions: Drug: ADVAIR DISKUS 250/50 mg BID
- Serevent 50 mcg BID (Active Comparator): Salmeterol xinafoate Inhalation Powder (SEREVENT DISKUS) is indicated for the long-term, twice-daily (morning and evening), administration in the maintenance treatment of bronchospasm associated with COPD (including emphysema and chronic bronchitis).
  Interventions: Drug: SEREVENT 50 mcg BID

INTERVENTIONS:
Drug: ADVAIR DISKUS 250/50 mg BID — Fluticasone propionate/salmeterol 250/50 mcg BID in the DISKUS formulation (ADVAIR DISKUS) is a combination product containing a corticosteroid and a long-acting beta2-adrenergic agonist, indicated in the US for the maintenance treatment of airflow obstruction and reducing exacerbations in patients with COPD.
  Other Names: FSC 250/50 mcg
  Arms: ADVAIR DISKUS 250/50 mcg BID
Drug: SEREVENT 50 mcg BID — Salmeterol xinafoate Inhalation Powder (SEREVENT DISKUS) is indicated for the long-term, twice-daily (morning and evening), administration in the maintenance treatment of bronchospasm associated with COPD (including emphysema and chronic bronchitis).
  Other Names: Salmeterol xinafoate 50 mcg
  Arms: Serevent 50 mcg BID

SUMMARY:
This trial is a randomized, double-blind, parallel-group, multicenter study to be conducted in the United States. The purpose of the study is to evaluate the rate of exacerbations of chronic obstructive pulmonary disease (COPD) following hospital discharge for an acute exacerbation of COPD, in patients receiving either fluticasone propionate/salmeterol combination product 250/50mcg BID or salmeterol 50mcg BID via DISKUS™ over 29 weeks. The study population will include patients hospitalized for an acute exacerbation of COPD. The target enrolment is 720 subjects at 80 study centers. The primary endpoint is the rate of exacerbation requiring hospitalization that occur more than 21 days post-discharge, emergency room visit or physician's office visit for an exacerbation of COPD requiring treatment with oral corticosteroids or oral corticosteroids and antibiotics. The secondary endpoint is the rate of COPD exacerbation requiring treatment with oral corticosteroids, antibiotics, and/or hospitalization (alone and in combination). Related efficacy endpoints include, time to first exacerbation of COPD requiring treatment with oral corticosteroids, antibiotics, and/or hospitalization (alone and in combination), pre-dose AM FEV1, the probability of premature withdrawal of subject from the study, and supplemental albuterol use, change in biomarkers of inflammation, including, surfactant protein D (SP-D), clara cell secretory protein 16 (CC-16) and high sensitivity C-reactive protein (hs-CRP). Health outcome assessments include domain scores evaluation for fatigue, dyspnea, emotional function and mastery, measured with the Chronic Respiratory Disease Questionnaire self-administered standardized format (CRQ-SAS); and symptoms (congestion, cough, phlegm, mucus, chest discomfort, shortness of breath and sleep disturbance), assessed by the EXAcerbations of Chronic pulmonary disease Tool (EXACT). Albuterol will be supplied to study subjects for use as-needed throughout the study. Safety will be assessed by monitoring of adverse events.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in this study must meet all of the following criteria:

* Male or female of at least 40 years of age at screening.

To be eligible for entry into the study, females of childbearing potential must commit to the consistent and correct use of an acceptable method of birth control starting on the day of visit 1, throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of six days), as defined by any one of the following:

* Abstinence Females of childbearing potential who are not sexually active must commit to complete abstinence from intercourse
* Oral contraceptive (either combined estrogen/progestin or progestin only)
* Injectable progestogen
* Implants of levonorgestrel or etonogestrel
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year,
* Male partner who is sterile (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study and is the sole sexual partner for that female subject, or
* Double-barrier method; condom or occlusive cap (diaphragm or cervical /vault caps) plus spermicide.
* Current or former smokers with a >10 pack-year cigarette smoking history [number of pack years = (number of cigarettes per day / 20) X number of years smoked (e.g., 10 pack-years is equal to 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years]. Former smokers are defined as those who have quit smoking for at least 3 months prior to the screening visit.
* Any of the following populations:
* Patients hospitalized for a duration not exceeding 10 days due to an acute exacerbation of COPD, and who must be randomized within 10 days post-discharge.
* Patients with COPD who were treated and held for observation in the emergency department (i.e. emergency room, ER) for at least 24 hours due to an acute exacerbation of COPD, and who must be randomized within 10 days post-discharge.
* Patients who received oral corticosteroids or oral corticosteroids and antibiotics for treatment of an exacerbation of COPD during a physician's office visit and who must be randomized within 10 days of the visit, and who have been hospitalized within the previous six months due to an acute exacerbation of COPD.
* Clinical diagnosis of COPD (for at least 6 months). The following definition of COPD from the American Thoracic Society (ATS) will be used: COPD is a disease state characterized by the presence of airflow obstruction due to chronic bronchitis or emphysema; the airflow obstruction is generally progressive, may be accompanied by airway hyper-reactivity, and may be partially reversible [American Thoracic Society, 1995].
* Documented evidence (within a year prior to Visit 1) in the medical chart of spirometry confirming the diagnosis of COPD and/or spirometry performed prior to randomization (Visit 2) that confirms pre-bronchodilator FEV1/FVC ratio less than or equal to 0.70 and pre-bronchodilator FEV1 <70% of predicted.
* Review and subject's completion of written informed consent: a subject-signed and dated written informed consent (form) must be obtained prior to any study procedure, and the subject must be willing to comply with all the requirements of the study protocol.
* Subject must be able to read, comprehend, and record information in English or Spanish.

Exclusion Criteria:

* Subjects meeting any of the following criteria must not be enrolled in the study:
* Diagnosis of pneumonia, congestive heart failure (CHF), or other complicating co-morbid condition while hospitalized within the last 6 months for an exacerbation of COPD.
* Historical or current evidence of clinically significant uncontrolled disease including, but not limited to, those listed below. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subjects at risk through study participation, or which would affect the safety analysis or other analyses if the disease/condition exacerbated during the study.
* A previous lung resection surgery (e.g. lobectomy, pneumonectomy, etc) within the year preceding Visit 1 (Screening)
* Asthma as primary diagnosis
* Lung cancer
* Cystic fibrosis, pulmonary fibrosis, active tuberculosis, or sarcoidosis
* Clinically significant cardiac arrhythmias
* Uncontrolled hypertension
* Unstable angina
* Current malignancy or a previous history of cancer in remission for < 5yrs (localized basal cell or squamous cell carcinoma of the skin that has been resected is not excluded)
* Uncontrolled diabetes mellitus
* Uncontrolled hyperthyroidism or hypothyroidism
* Immunologic compromise
* Cushing's or Addison's disease
* An abnormal 12-lead electrocardiogram (ECG) at Visit 1 (Screening) deemed to be clinically significant by the investigator.
* A chest X-ray or computed tomography (CT) scan performed in the 6 months preceding Visit 1 that revealed evidence of clinically significant abnormalities not believed to be due to the presence of COPD. If the subject does not have a record of a chest X-ray, one must be obtained and reviewed prior to randomization.
* Female patients with a positive urine pregnancy test at Visit 1.
* Any infirmity, physical disability, or geographic location that would limit compliance for scheduled visits.
* Any adverse reaction, immediate or delayed, hypersensitivity to any Beta-agonist, sympathomimetic drug, or corticosteroid including any components of the study drug formulations.
* Limited ability to provide a valid informed consent due to psychiatric disease, intellectual deficiency, poor motivation, current substance abuse (including illicit drugs and alcohol), or neurological disorders that might interfere with completion of study procedures or hearing problems that may impede effective communication.
* Study site staff (i.e. participating investigator, sub-investigator, study coordinator, employee of the participating investigator) or family members of site staffs.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 639 (Actual)
Dates: Start 2010-04-30; Primary Completion 2012-04-01 (Actual); Study Completion 2012-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (93):
- United States (69):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Florence, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Sepulveda, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Bay Pines, Florida
  - GSK Investigational Site, Brandon, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Kissimmee, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Belleville, Illinois
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Livonia, Michigan
  - GSK Investigational Site, Fridley, Minnesota
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, North Syracuse, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Elizabeth City, North Carolina
  - GSK Investigational Site, Statesville, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Fort Mill, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Seneca, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Spokane, Washington
- Argentina (18):
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, San Juan Bautista, Buenos Aires
  - GSK Investigational Site, Comodoro Rivadavia, Chubut Province
  - GSK Investigational Site, Concepción del Uruguay, Entre Ríos Province
  - GSK Investigational Site, Godoy Cruz, Mendoza Province
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Bariloche, Río Negro Province
  - GSK Investigational Site, Cipolletti, Río Negro Province
  - GSK Investigational Site, El Calafate, Santa Cruz Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Corrientes
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, San Salvador de Jujuy
  - GSK Investigational Site, Santa Fe
- Norway (6):
  - GSK Investigational Site, Bodø
  - GSK Investigational Site, Levanger
  - GSK Investigational Site, Stavanger
  - GSK Investigational Site, Trondheim
  - GSK Investigational Site, Tønsberg
  - GSK Investigational Site, Volda

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Ohar JA, Crater GD, Emmett A, Ferro TJ, Morris AN, Raphiou I, Sriram PS, Dransfield MT. Fluticasone propionate/salmeterol 250/50 mug versus salmeterol 50 mug after chronic obstructive pulmonary disease exacerbation. Respir Res. 2014 Sep 24;15(1):105. doi: 10.1186/s12931-014-0105-2. PMID 25248764
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 113874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113874 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- FSC 250/50: Participants (par.) self-administered Fluticasone Propionate/Salmeterol (FSC) combination product 250/50 micrograms (µg) twice daily (BID) (one inhalation in the morning and another inhalation in the evening, approximately 12 hours apart) for 29 weeks, approximately.
- SAL 50: Participants self-administered Salmeterol (SAL) 50 µg BID (one inhalation in the morning and another inhalation in the evening, approximately 12 hours apart) for 29 weeks, approximately.
Period: Overall Study
Arm/Group | FSC 250/50 | SAL 50
Started | 314 | 325
Completed | 208 | 204
Not Completed | 106 | 121
Not completed — Adverse Event | 28 | 28
Not completed — Withdrawal by Subject | 25 | 32
Not completed — Lack of Efficacy | 16 | 25
Not completed — Protocol Violation | 14 | 12
Not completed — Physician Decision | 13 | 17
Not completed — Lost to Follow-up | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- FSC 250/50: Participants self-administered Fluticasone Propionate/Salmeterol (FSC) combination product 250/50 micrograms (µg) twice daily (BID) (one inhalation in the morning and another inhalation in the evening, approximately 12 hours apart) for 29 weeks, approximately.
- Total: Total of all reporting groups
Arm/Group | FSC 250/50 | SAL 50 | Total
Number analyzed (Participants) | 314 | 325 | 639
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.1 (9.15) | 62.7 (9.30) | 62.9 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 151 | 291
  Male | 174 | 174 | 348
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage (AA/AH) | 26 | 22 | 48
  American Indian or Alaska Native | 1 | 2 | 3
  Asian-Japanese/South East and East Asian Heritage | 0 | 1 | 1
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 284 | 300 | 584
  AA/AH & American Indian or Alaska Native | 1 | 0 | 1
  American Indian or Alaska Native & White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Par. With Chronic Obstructive Pulmonary Disease (COPD) EXs Requiring Hospitalization That Occurred >21 Days Post-discharge/Physician's Office Visit for a COPD EX Requiring Treatment With Oral Corticosteroids (OCSs) or OCSs and Antibiotics (ABs)
Description: A COPD exacerbation (EX) was defined as the worsening of >=2 major symptoms (dyspnoea, sputum volume, sputum purulence [containing/discharging pus]) or the worsening of any 1 major symptom together with any 1 minor symptom (sore throat, cold [nasal discharge and/or nasal conjestion], fever without other cause, increased cough or wheeze) for at least 2 consecutive days. COPD EXs were identified by symptom review, and/or were based on investigator judgment (via phone contact or at a clinic visit). Hospitalization had to occur >21 days post-discharge/physician's office visit for a prior COPD EX.
Time Frame: From 21 days post-discharge (hospital or emergency room) or physician's office visit, up to 29 weeks
Population: Intent-to-Treat (ITT) Population: all participants randomized to study drug
Measure: Number; unit: participants
Arm/Group | FSC 250/50 | SAL 50
Number analyzed (Participants) | 314 | 325
participants | 43 | 39

2. Primary Outcome: Number of Participants With the Indicated Number of EXs of COPD Requiring Hospitalization That Occurred More Than 21 Days Post-discharge or Physician's Office Visit for an EX of COPD Requiring Treatment With OCSs or OCSs and ABs
Description: A COPD EX was defined as the worsening of >=2 major symptoms (dyspnoea, sputum volume, sputum purulence [containing/discharging pus]) or the worsening of any 1 major symptom together with any 1 minor symptom (sore throat, cold [nasal discharge and/or nasal conjestion], fever without other cause, increased cough or wheeze) for at least 2 consecutive days. COPD EXs were identified by symptom review, and/or were based on investigator judgment (via phone contact or at a clinic visit). Hospitalization had to occur more than 21 days post-discharge or physician's office visit for a prior COPD EX.
Time Frame: From 21 days post-discharge (hospital or emergency room) or physician's office visit, up to 29 weeks
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | FSC 250/50 | SAL 50
Number analyzed (Participants) | 314 | 325
participants
  0 | 271 | 286
  1 | 36 | 31
  2 | 7 | 5
  3 | 0 | 2
  4 | 0 | 1

3. Primary Outcome: Number of EXs of COPD Requiring Hospitalization That Occurred More Than 21 Days Post-discharge or Physician's Office Visit for an EX of COPD Requiring Treatment With OCSs or OCSs and ABs
Description: as for outcome 2
Time Frame: From 21 days post-discharge (hospital or emergency room) or physician's office visit, up to 29 weeks
Population: ITT Population. Only those participants with an EX requiring hospitalization were assessed.
Measure: Number; unit: Exacerbations
Arm/Group | FSC 250/50 | SAL 50
Number analyzed (Participants) | 43 | 39
Exacerbations | 50 | 51
Statistical Analysis 1: Comparison: FSC 250/50 vs SAL 50; Test type: Superiority or Other; p = 0.710, Negative bionomial regression model; Treatment comparison ratio = 0.917, 95% CI 2-sided [0.581 to 1.447] — Annualized rate estimates, the treatment comparison ratio, the confidence interval, and the p-value are from a negative binomial regression model with terms for treatment, country, randomization stratum, baseline severity, and time on treatment

4. Secondary Outcome: Number of Participants With an EX of COPD Requiring Treatment With OCSs, Treatment With ABs, and/or Hospitalization
Description: A COPD EX was defined as the worsening of >=2 major symptoms (dyspnoea, sputum volume, sputum purulence [containing/discharging pus]) or the worsening of any 1 major symptom together with any 1 minor symptom (sore throat, cold [nasal discharge and/or nasal conjestion], fever without other cause, increased cough or wheeze) for at least 2 consecutive days. COPD EXs were identified by symptom review, and/or were based on investigator judgment (via phone contact or at a clinic visit).
Time Frame: From Baseline up to Week 29, approximately
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | FSC 250/50 | SAL 50
Number analyzed (Participants) | 314 | 325
participants | 102 | 115

5. Secondary Outcome: Number of EXs of COPD Requiring Treatment With OCSs, Treatment With ABs, and/or Hospitalization (Alone and in Combination)
Description: as for outcome 4
Time Frame: From Baseline up to Week 29, approximately
Population: ITT Population. Only those participants with an EX were assessed for hospitalization, treatment with OCSs, and treatment with ABs.
Measure: Number; unit: exacerbations
Arm/Group | FSC 250/50 | SAL 50
Number analyzed (Participants) | 314 | 325
exacerbations
  Number of EXs, n=314,325 | 156 | 182
  Number of EXs requiring hospitalization, n=156,182 | 50 | 51
  Number of EXs treated with OCSs, n=156, 182 | 140 | 167
  Number of EXs treated with ABs, n=156, 182 | 121 | 144

ADVERSE EVENTS:
Arm/Group | FSC 250/50 | SAL 50
Serious Adverse Events (participants affected / at risk) | 75/314 | 82/325
Other Adverse Events (participants affected / at risk) | 88/314 | 105/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC 250/50 (N=314) | SAL 50 (N=325)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 47 | 51
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 5
Bronchitis (Infections and infestations) | 3 | 3
Cellulitis (Infections and infestations) | 2 | 1
Lobar pneumonia (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Sepsis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Encephalitis herpes (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Infective exacerbation, chronic obstructive airways disease (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 3
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Labile hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peritoneal carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FSC 250/50 (N=314) | SAL 50 (N=325)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 47 | 51
Headache (Nervous system disorders) | 19 | 19
Upper respiratory tract infection (Infections and infestations) | 15 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 13
Diarrhoea (Gastrointestinal disorders) | 11 | 10
Oedema peripheral (General disorders) | 6 | 14
Nausea (Gastrointestinal disorders) | 5 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.